CLINICAL TRIAL: NCT05905107
Title: Effects of Neurodynamic Sequencing on Pain, Wrist Range of Movement and Functional Disability in Patients With Carpal Tunnel Syndrome
Brief Title: Neurodynamic Sequencing in Patients With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC_FSD_00325
Record Dates: First submitted 2023-05-09; First posted 2023-06-15 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group A (Experimental): These patients will be treated by nerve sequencing proximal to distal in 3 sets of 15 repetitions in one session on alternate days for 4 weeks. For this, participants will be given a comfortable supine lying position. ULTT method will be implemented to the ipsilateral upper limb given in the table below
  Interventions: Other: Neurodynamic Slider Technique from Proximal to Distal
- Interventional Group B (Active Comparator): These patients will be treated by nerve sequencing distal to proximal in 3 sets of 10 repetitions in one session for 4 weeks. For this, participants will be given a comfortable supine lying position. ULTT method will be implemented to the ipsilateral upper limb
  Interventions: Other: Neurodynamic Slider Technique from Distal to Proximal

INTERVENTIONS:
Other: Neurodynamic Slider Technique from Proximal to Distal — Neurodynamic Slider Technique from proximal to distal at wrist, elbow and neck
  Arms: Interventional Group A
Other: Neurodynamic Slider Technique from Distal to Proximal — Neurodynamic Slider Technique from proximal to distal at wrist, elbow and neck
  Arms: Interventional Group B

SUMMARY:
Carpal tunnel syndrome is a compressive neuropathy of median nerve in the fascial tunnel at wrist which causes pain, numbness ,and tingling in the extremities. Common treatment options used in the treatment of carpal tunnel syndrome are conservative and surgical treatment option is better, this question is still a topic requiring more and more clinical trials. Neuromobilisation described by Butler is one of the treatment options which are used in the treatment of carpal tunnel syndrome in conjunction with other conservative measures.

This proposed study will find out the effectiveness of Neuromobilisation in treatment of carpal tunnel syndrome. As there is very little evidence available which Neuromobilisation technique is effective and what are the types of patients which can get benefit from this technique. This study will find out the effect of Neuromobilisation in patients suffering from carpal tunnel syndrome of non traumatic origin. This is a randomized clinical trial. Target population is patients suffering from carpal tunnel syndrome of non-traumatic origin. Data will be collected from District Headquarter Hospital Faisalabad. This study will include 56 participants according to the selection criteria. The participants will be randomly divided into two groups through sealed opaque envelop method.

Group A will recruit 28 patients which fulfill the inclusion criteria. These patients will be treated by nerve sequencing proximal to distal in 3 sets of 15 repetitions in one session on alternate days for 4 weeks. Group B will recruit 28 patients which fulfill the inclusion criteria. These patients will be treated by nerve sequencing distal to proximal in 3 sets of 10 repetitions in one session for 4 weeks. The Statistical analysis will be performed through SPSS Software 21.

ELIGIBILITY:
Inclusion Criteria:

* Patients positive for provocative test ( Phalen's test, Wrist decompression test and tinnel test).

Exclusion Criteria:

* Inflammation around the wrist
* Tumor around the wrist
* Rheumatoid Arthritis
* Osteoporosis
* Joint Hypermobility

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Pain at wrist joint | 4 weeks
  Pain will be assessed by using Numerical Pain Rating Scale Pain will be assessed by using Numerical Pain Rating Scale
Wrist Range of Movement at wrist joint | 4 weeks
  Range of motion will be assessed by using Goniometer
Functional Ability at wrist joint | 4 weeks
  Functional Ability will be assessed by using Boston Carpal tunnel syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Sahreen Anwar, Ph.D, Principal Investigator — Riphah International University
Locations (1):
- District Headquarters Hospital, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No